CLINICAL TRIAL: NCT04891367
Title: Cognitive Behavioral Group Treatment for Adolescents With Obsessive-compulsive Disorder: An Open Trial Benchmarking Against Individual Treatment Effectiveness and Quality of Life
Brief Title: Cognitive Behavioral Group Treatment for Obsessive-compulsive Disorder in Youth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Aarhus University Hospital (Other)
Collaborators: Jascha Fonden (Other); Region midtjyllands sundhedsvidenskabelige forskningsfond (Unknown); Sygekassernes Helsefond (Other); Region Midtjyllands Psykiatriske Forskningsfond (Unknown)
Responsible Party: Principal Investigator, Katja Anna Hybel, Senior researcher, PhD, Aarhus University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCBT OCD study - BUA
Record Dates: First submitted 2021-05-02; First posted 2021-05-18 (Actual); Last update posted 2022-09-27 (Actual); Status verified 2022-09

CONDITIONS: Obsessive-Compulsive Disorder; Cognitive Behavioral Therapy; Adolescent
Keywords: Cognitive behavioral Group Therapy; Youth; OCD
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group CBT (Experimental): Group cognitive behavioral therapy for obsessive compulsive disorder in youth
  Interventions: Other: Cognitive behavioral therapy

INTERVENTIONS:
Other: Cognitive behavioral therapy — The G-CBT manual for adolescents has been developed in the OCD-clinic in Aarhus and pilot tested in Aarhus. The G-CBT manual is based on the NordLOTS I-CBT manual in overall content and structure, with a few additional elements added with inspiration from previous individual and group CBT literature as well as the author's ideas. The main therapeutic ingredient is exposure and response prevention. The manual is made up of three individual family sessions, 13 weekly adolescent group sessions, three parent group sessions and two adolescent group booster sessions.The manual contains detailed guiding of therapists for each session and a comprehensive collection of working sheets for the adolescents to be used during sessions.

SUMMARY:
Obsessive-compulsive disorder (OCD) is a debilitating disorder characterized by unwanted intrusive thoughts and disrupting repetitive rituals. Epidemiological studies estimate the prevalence of impairing OCD to be between 0.5-3.0 % in pediatric populations. Although OCD in youth is associated with substantial distress and functional impairment, access to evidence-based psychosocial treatments is limited. This is largely due to the fact that few clinicians are trained in the delivery of evidence-based treatments, such as exposure-based cognitive-behavioral therapy (CBT). Therefore it is of great importance to develop treatment programs that utilize therapist resources in the most efficient way.

Exposure-based CBT delivered in the context of a group, rather than individually, is one such option. However, there are currently no evidence-based group OCD treatment manuals for youth available to clinicians in Denmark. Therefore this project addresses an important clinical need. We evaluate a group-based CBT protocol for the treatment of youth with OCD, benchmarking treatment outcomes against data from a previous trial evaluating individual-based CBT and by comparing outcomes against a short waiting list period. Further, we will explore the impact of group-based CBT over a 36-month open follow-up interval on general functioning, relapse, recurrence rates, and the need for other treatments. Finally, a brief youth questionnaire assessing overall symptom severity relevant for the evaluation of outcomes in pediatric OCD will be translated and validated for future clinical and research use in Denmark.

The project will include 72 adolescents with a primary diagnosis of OCD referred for assessment and treatment at the OCD Clinic at Department of Child and Adolescent Psychiatry, Aarhus University Hospital, Psychiatry, Denmark. For benchmarking of treatment outcomes, the project will compare the results from the group-based CBT with data from 45 Danish patients previously enrolled in the individual-based CBT of the Nordic Long Term OCD Treatment Study at the same clinic.

DETAILED DESCRIPTION:
Aims and hypotheses. The main objective of the present study is to develop a group delivered treatment manual for youth with OCD and evaluate its efficacy relative to (1) a waiting list control condition and (2) outcomes from existing data from a study of individually delivered CBT using a benchmarking strategy. The efficacy of the new treatment manual will be evaluated at the end of 13 weeks of acute treatment and at 3-, 6- , 12-, 24- and 36-month follow-up.

Based on the previous research we hypothesize that: (i) G-CBT will show superiority to the waiting period condition, and (ii) G-CBT will show similar effectiveness compared to I-CBT at the end of acute treatment as well as at longer-term follow-up assessment points.

Secondary aims are to evaluate predictors of treatment response to G-CBT and to identify specific response trajectories, i.e. patterns of symptom fluctuation during treatment.

Based on the previous literature we want to explore whether: (1) youth in families with higher levels of family conflict, parental blame and lower levels of cohesion will benefit less from treatment when compared to youth without these family characteristics, (2) lower levels of initial and intermediate treatment motivation will be associated with lower levels of treatment gains, and (3) specific patient response trajectories possibly associated with the onset of specific treatment ingredients (i.e., initial psychoeducation, in session exposure and response prevention, specific work on obsessions, work meetings with parents, etc.) and/or with patient characteristics, i.e. OCD subtypes, can be identified.

Further, the aim is to develop and/or evaluate relevant Danish versions of clinical instruments for the assessment of pediatric OCD (symptoms and severity). More specifically, one aim is to develop and evaluate a short self-rating of OCD severity for youth with OCD, which can be utilized by therapists during treatment and as a tool for youth's self-monitoring of symptoms.

Procedures. Eligible patients will be recruited as they are consecutively referred to the OCD Clinic at Department of Child and Adolescent Psychiatry, Aarhus University Hospital, Psychiatry, Denmark.

Seventy-two adolescents, 13-17 years old will be included in the study, corresponding to inclusion of approximately 140 adolescents into twenty treatment groups.

The benchmarking sample includes all 13- to 17-year-old Danish participants from the aforementioned Scandinavian pediatric multicenter OCD CBT study, NordLOTS. NordLOTS data provide a unique opportunity to benchmark outcomes from the two different CBT formats delivered at the same clinic. Therefore, the procedures used in the present study are largely similar to the procedures used in NordLOTS (the Committee of Ethical Science file number: 20070140). Patients for the current study will be included as they are consecutively referred to the OCD Clinic and enrolled in the standard clinical assessment and treatment procedures. All assessments will be conducted by experienced external clinician raters (i.e., clinicians from the clinic who are not acting as therapists in the treatment of the assessed patient).

In order to be able to adjust data analyses for possible interdependence of observations due to group membership, patients who are offered G-CBT treatment (i.e. offered G-CBT as a part of the standard clinical procedures) but fall for study exclusion criteria (e.g. previously or presently treated with SSRI's) or patients who do not wish to participate in the extended assessment procedures in the project (i.e. decline participation after presented with project information at the first visit to the clinic) will be asked permission to use the following clinical data according to their clinical record: gender, age, age at OCD-onset, present psychiatric diagnoses, and CY-BOCS scores at pre-treatment, mid-treatment, end of acute treatment, and at 3 months follow-up.

Intervention The G-CBT manual for adolescents has been developed in the OCD-clinic in Aarhus and pilot tested in Aarhus and subsequently in collaboration with clinicians at the OCD Clinic, Queen Silvia Children's Hospital, Sahlgrenska University Hospital, Department of Child and Adolescent Psychiatry Gothenburg, Sweden, who also participated in NordLOTS. The G-CBT manual is based on the NordLOTS I-CBT manual63 in overall content and structure, with a few additional elements added with inspiration from previous individual and group CBT literature12,13,64-67 as well as the author's ideas. The NordLOTS manual is primarily based on a neurobiological model for psychoeducation, and the main therapeutic ingredient is exposure and response prevention. The additional or slightly altered elements in the G-CBT manual include: a) a stronger emphasis on cognitive aspects and goal-setting, b) introduction of formalized supportive "work-meetings" between children/adolescents and parents, c) exercises in thought focus strategies, d) verbalization of parents' recognition of the young patient's work and efforts during the program by a parent speech at the final treatment session, and e) introduction of an OCD farewell letter during the booster sessions. The number of individual family and parent sessions is largely modeled after the Australian OCD Busters manual (albeit, only the published journal paper reporting of this manual was available at the time of the development of the Danish manual)13. The manual is made up of three individual family sessions, 13 weekly adolescent group sessions, three parent group sessions and two adolescent group booster sessions conducted after one and three months. The adolescent group sessions are conducted by two therapists and the parent group sessions are conducted by one therapist. The manual contains detailed guiding of therapists for each session and a comprehensive collection of working sheets for the adolescents to be used during sessions.

Reliability of primary outcome measures and treatment fidelity ratings Following the previous procedures from NordLOTS, reliability ratings of primary outcome assessment will be performed by experienced clinicians on a random sample of 15 % of baseline and week 13 CY-BOCS interviews. All interviews will be videotaped and uploaded to the research database (RedCAP). An adaptation of the NordLOTS Treatment Integrity Scale (TIS)9 will be used to evaluate therapist fidelity to the CBT sessions. All therapy sessions will be videotaped and uploaded to the research database (RedCAP). A random sample of 15 % of all sessions will be scored by experienced semi-independent clinicians. In TIS 3 categories of treatment fidelity are evaluated on a four-point scale ranging from 1 = very poor compliance to 4 = very good compliance: (1) manual adherence, (2) competence in manual delivery, and (3) therapist relational competencies.

Power calculation and statistical analyses In total, we expect to include 72 experimental subjects treated with G-CBT and 45 subjects previously included in NordLOTS treated with I-CBT and completing the program. With reference to NordLOTS we expect a drop-out rate of 10 % during treatment9 and a further 12.5 % drop-out during the one-year post-treatment follow-up period. One-year Outcome for Responders of Cognitive Behavior Therapy for Child and Adolescent Obsessive-Compulsive Disorder.). Expected distribution, standard deviation and differences in response between waiting period condition and CBT calculated based on data from two previous studies showing CY-BOCS change scores of -1.09 (SD = 4.86) and 13.2 (SD = 6.41) respectively, indicates that the response within each subject group is normally distributed with a standard deviation of 5.69 and a change score mean difference between conditions of 14.29. If this mean difference between conditions holds true for the planned study we will be able to reject the null hypothesis i.e. that the means of the two conditions are equal with a probability (power) of 1.000 and a type I error probability of 0.05.

Descriptive statistics for sample characteristics as well as outcome measures will be calculated. In order to assess treatment effect, a multilevel linear mixed model with CY-BOCS severity score as primary outcome dependent variable including random slopes and intercept will be applied. To estimate the treatment effect measured with the CGI-S, a generalized linear effects model will be used. Waiting period vs. treatment condition CY-BOCS change scores will be estimated using a random effects model in order to adjust for differences in exposure length in the two conditions. Secondary outcome measures include KINDL, OBQ-CV, COIS, MFQ, and SCARED.

Out of the 269 patients in NordLOTS, the Aarhus site included 80. Of these, 45 were adolescents between the age of 13-17. The expected inclusion of 72 adolescents in the current study will be sufficient for comparative benchmarking and predictor analyses.

In the benchmarking analyses participant baseline demographics (age, gender, BQ), clinical characteristics (CY-BOCS, CGI, KINDL, C-GAS, CBCL, FAS, COIS, MFQ, SCARED, ASSQ) and scores on outcome measures (primary measures: CY-BOCS, CGI, KINDL; secondary measures: C-GAS, COIS, MFQ, SCARED, OBQ-CV) will be compared between the two samples using independent samples t-tests and Fisher's exact test. In order to adjust for possible interdependence of observations due to group membership, intra-class correlation coefficients (ICCs) will be calculated for primary outcome measures (CY-BOCS): ICC = (MSbetweengroup - MSwithingroup)/(MSbetweengroup + [n - 1] MSwithingroup). Pre- to post CY-BOCS change will be estimated as pre-post effect sizes [ES] where the ES equals the mean difference between pre-treatment and post-treatment scores divided by the standard deviation of the mean difference, adjusted by the correlation between the pre- and post-scores. Difference between the two interventions will be estimated by calculating the standardized mean difference between the pre-post change scores of the two samples, divided by a pooled estimate of the post-test standard deviations. Analyses will use an intention-to-treat (ITT) approach. A two-sample t-test for proportions will be conducted in order to examine the difference in participant completion rate between the current study and the benchmark study.

ELIGIBILITY:
Inclusion Criteria:

* 13 to 17 years of age
* A primary diagnosis of OCD according to Schedule for Affective Disorders and Schizophrenia for School-Age Children - Present and Lifetime version for DSM-IV (K-SADS-PL).
* Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS)24 total score ≥ 16.

Exclusion Criteria:

* meet the criteria for an intellectual disability (IQ < 70),
* meet the criteria for psychotic disorder according to DSM-5,
* meet the criteria for Asperger's, or Autistic syndrome with a Clinical Global Impression Scale - Severity (CGI-S) rating ≥ 4 or same or higher rating than CGI-S for OCD
* meet the criteria for PDD-NOS with a Clinical Global Impression Scale - Severity (CGI-S) rating ≥ 4 or same or higher rating than CGI-S for OCD
* meet the criteria for any co-occurring mental disorder according to the Diagnostic and statistical manual of mental disorders (DSM-5) with a CGI-S rating higher than CGI-S for OCD, indicating that OCD is not the primary treatment priority
* have been treated with CBT six months prior to inclusion,
* have been treated with (S)SRIs six months prior to inclusion (dose ≥50 mg),
* have inadequate Danish language proficiency or both parents have inadequate Danish language proficiency

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2017-08-15 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
The Children's Yale-Brown Obsessive Compulsive Scale | Pre-waiting period of 2-16 weeks/pre-treatment
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) 24 is a clinician rated, semi structured interview assessing past and current OCD symptom presentation as well as present OCD severity in patients aged 6-17 years. The instrument has a 72-item symptom checklist followed by 10 severity items, five for obsessions and five for compulsions (i.e., time occupied by symptoms, interference, distress, resistance, and degree of control over symptoms), with a total severity score ranging from 0 to 40. Higher scores indicate worse outcome. The instrument is the most frequently used to assess OCD in children and adolescents.
The Children's Yale-Brown Obsessive Compulsive Scale | Post-waiting period of 2-16 weeks/pre-treatment (within 2 weeks before the first group session)
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) 24 is a clinician rated, semi structured interview assessing past and current OCD symptom presentation as well as present OCD severity in patients aged 6-17 years. The instrument has a 72-item symptom checklist followed by 10 severity items, five for obsessions and five for compulsions (i.e., time occupied by symptoms, interference, distress, resistance, and degree of control over symptoms), with a total severity score ranging from 0 to 40. Higher scores indicate worse outcome. The instrument is the most frequently used to assess OCD in children and adolescents.
The Children's Yale-Brown Obsessive Compulsive Scale | Mid-intensive-treatment (between session 7 and 8 in the intensive treatment period)
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) 24 is a clinician rated, semi structured interview assessing past and current OCD symptom presentation as well as present OCD severity in patients aged 6-17 years. The instrument has a 72-item symptom checklist followed by 10 severity items, five for obsessions and five for compulsions (i.e., time occupied by symptoms, interference, distress, resistance, and degree of control over symptoms), with a total severity score ranging from 0 to 40. Higher scores indicate worse outcome. The instrument is the most frequently used to assess OCD in children and adolescents.
The Children's Yale-Brown Obsessive Compulsive Scale | Post-intensive-treatment (at termination of intensive treatment)
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) 24 is a clinician rated, semi structured interview assessing past and current OCD symptom presentation as well as present OCD severity in patients aged 6-17 years. The instrument has a 72-item symptom checklist followed by 10 severity items, five for obsessions and five for compulsions (i.e., time occupied by symptoms, interference, distress, resistance, and degree of control over symptoms), with a total severity score ranging from 0 to 40. Higher scores indicate worse outcome. The instrument is the most frequently used to assess OCD in children and adolescents.
The Children's Yale-Brown Obsessive Compulsive Scale | Post-booster-treatment (at termination of booster treatment - 3 months after the last session in the intensive treatment period)
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) 24 is a clinician rated, semi structured interview assessing past and current OCD symptom presentation as well as present OCD severity in patients aged 6-17 years. The instrument has a 72-item symptom checklist followed by 10 severity items, five for obsessions and five for compulsions (i.e., time occupied by symptoms, interference, distress, resistance, and degree of control over symptoms), with a total severity score ranging from 0 to 40. Higher scores indicate worse outcome. The instrument is the most frequently used to assess OCD in children and adolescents.
The Children's Yale-Brown Obsessive Compulsive Scale | 6 months follow-up
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) 24 is a clinician rated, semi structured interview assessing past and current OCD symptom presentation as well as present OCD severity in patients aged 6-17 years. The instrument has a 72-item symptom checklist followed by 10 severity items, five for obsessions and five for compulsions (i.e., time occupied by symptoms, interference, distress, resistance, and degree of control over symptoms), with a total severity score ranging from 0 to 40. Higher scores indicate worse outcome. The instrument is the most frequently used to assess OCD in children and adolescents.
The Children's Yale-Brown Obsessive Compulsive Scale | 12 months follow-up
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) 24 is a clinician rated, semi structured interview assessing past and current OCD symptom presentation as well as present OCD severity in patients aged 6-17 years. The instrument has a 72-item symptom checklist followed by 10 severity items, five for obsessions and five for compulsions (i.e., time occupied by symptoms, interference, distress, resistance, and degree of control over symptoms), with a total severity score ranging from 0 to 40. Higher scores indicate worse outcome. The instrument is the most frequently used to assess OCD in children and adolescents.
The Children's Yale-Brown Obsessive Compulsive Scale | 24 months follow-up
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) 24 is a clinician rated, semi structured interview assessing past and current OCD symptom presentation as well as present OCD severity in patients aged 6-17 years. The instrument has a 72-item symptom checklist followed by 10 severity items, five for obsessions and five for compulsions (i.e., time occupied by symptoms, interference, distress, resistance, and degree of control over symptoms), with a total severity score ranging from 0 to 40. Higher scores indicate worse outcome. The instrument is the most frequently used to assess OCD in children and adolescents.
The Children's Yale-Brown Obsessive Compulsive Scale | 36 months follow-up
  The Children's Yale-Brown Obsessive Compulsive Scale (CY-BOCS) 24 is a clinician rated, semi structured interview assessing past and current OCD symptom presentation as well as present OCD severity in patients aged 6-17 years. The instrument has a 72-item symptom checklist followed by 10 severity items, five for obsessions and five for compulsions (i.e., time occupied by symptoms, interference, distress, resistance, and degree of control over symptoms), with a total severity score ranging from 0 to 40. Higher scores indicate worse outcome. The instrument is the most frequently used to assess OCD in children and adolescents.
The Health-Related Quality of Life in children and adolescents - revised | Pre-waiting period of 2-16 weeks/pre-treatment
  The Health-Related Quality of Life in children and adolescents - revised (KINDL-R) measure key aspects of health related quality of life in children and adolescents. Separate questionnaires for ages 7-13 and 14-17 exist. A translated Danish version of the KINDL is available. This scale provides a more general evaluation of the young patient's overall well-being and thriving in several life areas: physical, emotional, self-esteem, family, friends, and school, representing the child's experiences during the past week. Each item is rated on a five-point Likert scale and all scores are transformed to a scale ranging from 0 to 100. All subscale scores are added together to form a total score, with higher scores indicating better outcome. The questionnaire has a disorder-related subscale that reflects the child's experience of OCD-related burden and this is not part of the total score. The primary outcome used in the present study is the KINDL-R self-report total score.
The Health-Related Quality of Life in children and adolescents - revised | Post-waiting period of 2-16 weeks/pre-treatment (within 2 weeks before the first group session)
  The Health-Related Quality of Life in children and adolescents - revised (KINDL-R) measure key aspects of health related quality of life in children and adolescents. Separate questionnaires for ages 7-13 and 14-17 exist. A translated Danish version of the KINDL is available. This scale provides a more general evaluation of the young patient's overall well-being and thriving in several life areas: physical, emotional, self-esteem, family, friends, and school, representing the child's experiences during the past week. Each item is rated on a five-point Likert scale and all scores are transformed to a scale ranging from 0 to 100. All subscale scores are added together to form a total score, with higher scores indicating better outcome. The questionnaire has a disorder-related subscale that reflects the child's experience of OCD-related burden and this is not part of the total score. The primary outcome used in the present study is the KINDL-R self-report total score.
The Health-Related Quality of Life in children and adolescents - revised | Mid-intensive-treatment (between session 7 and 8 in the intensive treatment period)
  The Health-Related Quality of Life in children and adolescents - revised (KINDL-R) measure key aspects of health related quality of life in children and adolescents. Separate questionnaires for ages 7-13 and 14-17 exist. A translated Danish version of the KINDL is available. This scale provides a more general evaluation of the young patient's overall well-being and thriving in several life areas: physical, emotional, self-esteem, family, friends, and school, representing the child's experiences during the past week. Each item is rated on a five-point Likert scale and all scores are transformed to a scale ranging from 0 to 100. All subscale scores are added together to form a total score, with higher scores indicating better outcome. The questionnaire has a disorder-related subscale that reflects the child's experience of OCD-related burden and this is not part of the total score. The primary outcome used in the present study is the KINDL-R self-report total score.
The Health-Related Quality of Life in children and adolescents - revised | Post-intensive-treatment (at termination of intensive treatment)
  The Health-Related Quality of Life in children and adolescents - revised (KINDL-R) measure key aspects of health related quality of life in children and adolescents. Separate questionnaires for ages 7-13 and 14-17 exist. A translated Danish version of the KINDL is available. This scale provides a more general evaluation of the young patient's overall well-being and thriving in several life areas: physical, emotional, self-esteem, family, friends, and school, representing the child's experiences during the past week. Each item is rated on a five-point Likert scale and all scores are transformed to a scale ranging from 0 to 100. All subscale scores are added together to form a total score, with higher scores indicating better outcome. The questionnaire has a disorder-related subscale that reflects the child's experience of OCD-related burden and this is not part of the total score. The primary outcome used in the present study is the KINDL-R self-report total score.
The Health-Related Quality of Life in children and adolescents - revised | Post-booster-treatment (at termination of booster treatment - 3 months after the last session in the intensive treatment period)
  The Health-Related Quality of Life in children and adolescents - revised (KINDL-R) measure key aspects of health related quality of life in children and adolescents. Separate questionnaires for ages 7-13 and 14-17 exist. A translated Danish version of the KINDL is available. This scale provides a more general evaluation of the young patient's overall well-being and thriving in several life areas: physical, emotional, self-esteem, family, friends, and school, representing the child's experiences during the past week. Each item is rated on a five-point Likert scale and all scores are transformed to a scale ranging from 0 to 100. All subscale scores are added together to form a total score, with higher scores indicating better outcome. The questionnaire has a disorder-related subscale that reflects the child's experience of OCD-related burden and this is not part of the total score. The primary outcome used in the present study is the KINDL-R self-report total score.
The Health-Related Quality of Life in children and adolescents - revised | 6 months follow-up
  The Health-Related Quality of Life in children and adolescents - revised (KINDL-R) measure key aspects of health related quality of life in children and adolescents. Separate questionnaires for ages 7-13 and 14-17 exist. A translated Danish version of the KINDL is available. This scale provides a more general evaluation of the young patient's overall well-being and thriving in several life areas: physical, emotional, self-esteem, family, friends, and school, representing the child's experiences during the past week. Each item is rated on a five-point Likert scale and all scores are transformed to a scale ranging from 0 to 100. All subscale scores are added together to form a total score, with higher scores indicating better outcome. The questionnaire has a disorder-related subscale that reflects the child's experience of OCD-related burden and this is not part of the total score. The primary outcome used in the present study is the KINDL-R self-report total score.
The Health-Related Quality of Life in children and adolescents - revised | 12 months follow-up
  The Health-Related Quality of Life in children and adolescents - revised (KINDL-R) measure key aspects of health related quality of life in children and adolescents. Separate questionnaires for ages 7-13 and 14-17 exist. A translated Danish version of the KINDL is available. This scale provides a more general evaluation of the young patient's overall well-being and thriving in several life areas: physical, emotional, self-esteem, family, friends, and school, representing the child's experiences during the past week. Each item is rated on a five-point Likert scale and all scores are transformed to a scale ranging from 0 to 100. All subscale scores are added together to form a total score, with higher scores indicating better outcome. The questionnaire has a disorder-related subscale that reflects the child's experience of OCD-related burden and this is not part of the total score. The primary outcome used in the present study is the KINDL-R self-report total score.
The Health-Related Quality of Life in children and adolescents - revised | 24 months follow-up
  The Health-Related Quality of Life in children and adolescents - revised (KINDL-R) measure key aspects of health related quality of life in children and adolescents. Separate questionnaires for ages 7-13 and 14-17 exist. A translated Danish version of the KINDL is available. This scale provides a more general evaluation of the young patient's overall well-being and thriving in several life areas: physical, emotional, self-esteem, family, friends, and school, representing the child's experiences during the past week. Each item is rated on a five-point Likert scale and all scores are transformed to a scale ranging from 0 to 100. All subscale scores are added together to form a total score, with higher scores indicating better outcome. The questionnaire has a disorder-related subscale that reflects the child's experience of OCD-related burden and this is not part of the total score. The primary outcome used in the present study is the KINDL-R self-report total score.
The Health-Related Quality of Life in children and adolescents - revised | 36 months follow-up
  The Health-Related Quality of Life in children and adolescents - revised (KINDL-R) measure key aspects of health related quality of life in children and adolescents. Separate questionnaires for ages 7-13 and 14-17 exist. A translated Danish version of the KINDL is available. This scale provides a more general evaluation of the young patient's overall well-being and thriving in several life areas: physical, emotional, self-esteem, family, friends, and school, representing the child's experiences during the past week. Each item is rated on a five-point Likert scale and all scores are transformed to a scale ranging from 0 to 100. All subscale scores are added together to form a total score, with higher scores indicating better outcome. The questionnaire has a disorder-related subscale that reflects the child's experience of OCD-related burden and this is not part of the total score. The primary outcome used in the present study is the KINDL-R self-report total score.

SECONDARY OUTCOMES:
The Clinical Global Impression Scale | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Clinical Global Impression Scale (CGI) is a brief clinician-rated scale that assess the overall severity and impact of symptoms. The score range from 0 to 6 and higher scores indicate worse outcome.
The Children's Global Assessment Scale | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Children's Global Assessment Scale (CGAS) is a single-item instrument rated on a 0 to 100-point scale that assesses overall impairment and functional strain, including all possible stressors in the daily life of the patient. Higher scores indicate worse outcome.
The Child Obsessive Compulsive Impact Scale - Child and Parent Versions - Revised (COIS-R-C/P) | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Child Obsessive Compulsive Impact Scale - Child and Parent Versions - Revised (COIS-R-C/P) assess the impact of OCD symptoms on the psychosocial functioning of the youth in the home, in social settings, and academic settings. The scale has 33 items rated on a four-point scale. The total scale scores range between 0 and 99 and higher scores indicate worse outcome.
The Screen for Child Anxiety Related Emotional Disorders | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Screen for Child Anxiety Related Emotional Disorders (SCARED - parent and child versions) assess symptoms of anxiety based on the DSM-IV. The scale has 41 items rated on a three-point scale. The total scale scores range from 0 to 82 and higher scores indicate worse outcome.
The Mood and Feelings Questionnaire | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Mood and Feelings Questionnaire (MFQ) assesses depressive symptoms. It has 13 items rated on a three-point scale. The total scale scores range from 0 to 26 and higher scores indicate worse outcome.
The Family Accommodation Scale | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Family Accommodation Scale (FAS) is a 12-item scale that assesses the family's accommodation to the child's OCD symptoms including the provision of reassurance or objects needed for compulsions, decreased behavioral expectations of the child, modification of family activities or routines, or assisting with avoidance. The total scale scores range from 12 to 48 and higher scores indicate worse outcome.

OTHER OUTCOMES:
The Obsessive Beliefs Questionnaire - child version | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Obsessive Beliefs Questionnaire - Child Version (OBQ-CV) evaluates cognitions in childhood OCD. The scale has 44 items rated on a five point Likert scale and is validated in children and adolescents aged 8 - 17.The OBQ-CV has previously been translated into Danish following standard translation back-translation procedures by the first author of this protocol in collaboration with one of the original authors (Ingrid Söchting, PhD) and the psychometric properties of the Danish version have been evaluated. The total scale scores range from 44 to 220 and higher scores indicate worse outcome.
The Obsessive Compulsive Inventory - child version | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Obsessive Compulsive Inventory - child version (OCI-CV) is a well-established 21-item questionnaire assessing the frequency of obsessions and compulsions commonly present in OCD. The scale is suited to children and adolescents 7 - 17 years of age and has items covering seven symptom subtypes: washing, checking, hoarding, doubting, ordering, obsessing and neutralizing, and each item is scored on a three-point scale. The psychometric properties of the OCI-CV has been evaluated in several clinical samples as well as a large non-clinical sample. The scale has been translated for this study according to state-of-the art translation back-translation methods. The total scale scores range from 0 to 22 and higher scores indicate worse outcome.
The Mini Youth OCD Scale | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Mini Youth OCD Scale (MYOCD) assess overall OCD severity rated by the youth. The instrument is developed for this study by three of the authors of the present protocol. The scale has seven questions: three regarding severity (time spent on symptoms, interference in daily life activities, and level of perceived distress by symptoms), two regarding resistance (perceived effort in resistance to symptoms, and perceived control when resisting symptoms), one concerning avoidance behavior, and one reflecting the patient's perception of overall OCD severity. Prior to rating of the seven items the youth is asked to note the five most severe symptoms during the last week. The overall severity scale scores range from 0 to 4 and higher scores indicate worse outcome.
The Family Environment Scale | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Family Environment Scale (FES) assesses the social functioning of the family. The scale has 90 items rated either true or false. The subscales tapping level of conflict and cohesion will be applied in the present study. The total scale scores range from 0 to 90 and higher scores indicate worse outcome.
The Parental Attitudes and Behaviors Scale | Pre-wait/pre-treatment; Post-wait/pre-treatment; Mid-intensive-treatment; Post-intensive-treatment; Post-booster-treatment; 6 months follow-up; 12 months follow-up; 24 months follow-up; 36 months follow-up
  The Parental Attitudes and Behaviors Scale (PABS) is a 22-item scale evaluating how parents perceive their children's OCD symptoms as well as their parenting behavior in relation to OCD. The scale consists of the three sub-scales: Blame, Accommodation, and Empowerment. The total scale scores range from 22 to 110 and higher scores indicate worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Katja A Hybel, PhD, Principal Investigator — Aarhus University Hospital, Psychiatry, Department of Child and Adolescent Psychiatry
Locations (1):
- Katja Anna Hybel, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No